CLINICAL TRIAL: NCT06147739
Title: Evaluation Treatment Outcomes of Anterior Open Bite Treated With Maxillary Intrusive Force by Temporary Anchorage Devices
Brief Title: Evaluation Treatment Outcomes of Anterior Open Bite Treated by Temporary Anchorage Devices
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Bayan Saaidi, Principal Investigator Dr. Baian Msaaid Saaidi, Faculty of Dental Medicine for Girls
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORTHO-109-2-G
Record Dates: First submitted 2023-11-12; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Anterior Openbite Malocclusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Temporary Anchorage Devices — intrusion

SUMMARY:
The present study will be performed to Evaluate the treatment outcome of anterior open bite by temporary anchorage device on buccal and palatal mini screws

ELIGIBILITY:
Inclusion Criteria:

1. Patients age range 13-18 years old.
2. Patients have anterior open bite.
3. Normal healthy patient.
4. Patient have healthy oral tissues.
5. Patient have class I or II jaw relationship.
6. Patient have complete set of permanent teeth except the wisdom tooth.

Exclusion Criteria:

1. Uncooperative patient and parents.
2. patient who had undergo previous orthodontic treatment.
3. Patient with class III jaw relationship.

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-08-11 (Actual); Primary Completion 2023-12-11 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
open bite closure | 1 year
  the change in amount of open bite detected by mm. which measured from the cast model and from cephalometric x ray.

CONTACTS AND LOCATIONS:
Locations (1):
- Alazhar, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-16): https://cdn.clinicaltrials.gov/large-docs/39/NCT06147739/Prot_SAP_000.pdf